CLINICAL TRIAL: NCT04695717
Title: The Extensive, Double-blind, Randomized, Placebo-controlled Phase 3 Study to Evaluate the Safety and Immunogenicity of the Seasonal Inactivated, Split Virion, Trivalent Influenza Vaccine (IVACFLU-S) Produced in Children and the Elderly in Vietnam
Brief Title: This Study Was Conducted to Evaluate the Safety and Immunogenicity of IVACFLU-S Produced in Children From 6 Months to Under 18 Years Old and the Elderly Over 60 Years Old in Vietnam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vietnam Military Medical University (Other)
Collaborators: Institute of Vaccines and Medical Biologicals, Vietnam (Industry); Vietstar Biomedical Research (Industry)
Responsible Party: Principal Investigator, Pham Ngoc Hung, Principal Investigator, Vietnam Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VX.2020.01
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Influenza
Keywords: Influenza; vaccine; Seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Placebo Comparator): Received two doses of IVACFLU-S vaccine intramuscularly in children aged 6 months to under 9 years old and one dose of IVACFLU-S vaccine in children from 9 years old to under 18 years old adult over 60 years old
  Interventions: Biological: IVACFLU-S
- Placebo (Other): Received two doses of placebo intramuscularly in children aged 6 months to under 9 years old and one dose placebo in children from 9 years old to under 18 years old adult over 60 years old
  Interventions: Biological: IVACFLU-S

INTERVENTIONS:
Biological: IVACFLU-S — The Seasonal Inactivated, Split Virion, Trivalent Influenza Vaccine (TIV) were purified by the method of super centrifugation to create gradient segments in sucrose sugar produced by IVAC, or placebo produced by IVAC. Vaccines are produced on eggs, inactivated with formaldehyde. The dose of the vaccine tested was 15 mcg of HA for each antigen component in 0.5 ml.
  The influenza virus strains used to produce the 2020-2021 seasonal vaccine will also be provided by the NIBSC, which will be used according to WHO's recommendation, which is expected to include the following Southern Hemisphere strains:
  Influenza A / H1N1 strain: Recombinant strain IVR-190 44250 E12 of the strain (A / Brisbane / 02/2018).
  Influenza strain A / H3N2: strain IVR-197 (H3N2) 44850 E14 recombinant strain (A / South Australia / 34/2019).
  Flu strain B (B / Washington / February 2019).

SUMMARY:
This was an extensive, double-blind, randomized, placebo-controlled phase 3 study that aimed to evaluate the safety and immunogenicity of the seasonal inactivated, split virion, trivalent influenza vaccine (IVACFLU-S) in children from 6 months to under 18 years old and the elderly over 60 years old in Vietnam.

The main target:

Evaluating the safety of the single or double dose of seasonal influenza vaccine (IVACFLU-S) in Vietnamese children aged 6 months to 17 years and adults over 60 years old.

Evaluating the immunogenicity of the seasonal inactivated, split virion, trivalent influenza vaccine (IVACFLU-S) after 1st injection on day 22 (+7) for groups ≥ 9 years old or day 49 (+7) for groups of 6 months to 8 years for each antigenic component of the vaccine.

DETAILED DESCRIPTION:
The seasonal inactivated, split virion, trivalent influenza vaccine (TIV) were purified by the method of super centrifugation to create gradient segments in sucrose sugar produced by IVAC, or placebo produced by IVAC. Vaccines are produced on eggs, inactivated with formaldehyde. The dose of the vaccine tested was 15 mcg of HA for each antigen component in 0.5 ml. The influenza virus strains used to produce the 2020-2021 seasonal vaccine will also be provided by the NIBSC, which will be used according to WHO recommendations, which are expected to include the following Southern Hemisphere strains:

Influenza A / H1N1 strain: Recombinant strain IVR-190 44250 E12 of the strain (A / Brisbane / 02/2018).

Influenza strain A / H3N2: strain IVR-197 (H3N2) 44850 E14 recombinant strain (A / South Australia / 34/2019).

Flu strain B (B / Washington / February 2019). Extensive phase 3 was conducted 2 sites: District Health Center (DHC) of Vu Thu, Thai Binh, Vietnam; and DHC of Binh Luc, Ha Nam. Subjects were from two age groups: 6 months-under 18 years and over 60 years. Both safety and immunogenicity were assessed

ELIGIBILITY:
Inclusion Criteria:

*Groups from 6 months to under 18 years:

* Must have a sponsor (Father / Mother / Legal relative) and get the consent of the sponsor by signing a consent form to participate in the study. (Groups from 6 months to 8 years old must have a direct sponsor, groups 9-17 years old must have an indirect sponsor).
* The sponsor must be able to read and write and must commit to taking the child or asking the child to visit on schedule.
* If the Sponsor is not the child's parent, he/she must get the consent of the child's father/mother in writing.
* Healthy or previous acute illness but stabilized within 2 weeks before injection.
* No chronic disease (cancer, heart failure, kidney, liver ...) or chronic disease that has stabilized 3 months before injection.
* Children under 1 year old: Must have gestational age ≥ 37 and ≤ 42 weeks at birth and birth weight> 2500g and not have congenital disease.

Children <60 months of age are not severely malnourished (not exceeding I) Children 6 months to 8 years old who have never received a seasonal flu vaccine (from birth).

* Female adolescents who are likely to become pregnant need to be informed of possible risks to the fetus if participating in the study and if participating in the study, must comply with contraceptive measures during the period. research.

  *Group over 60 years old
* Can read, write (self-report) and ready to sign the consent form to participate in research.
* Ability to participate in scheduled visits and adhere to all procedures of testing.
* Be healthy or have a stable medical condition through history exploitation and physical examination. For subjects who have medical problems or symptoms/signs, the medical problems or symptoms/signs must be consistently controlled or unchanged within the past 3 months. If you are using medication to treat that medical problem, the dose should be stable for at least 1 month before the product is injected.
* For female subjects who are still fertile:

Are not breastfeeding, or are not pregnant (based on a negative urine test) and are not planning to become pregnant until Day 22. For women who have not had sterilization surgery (hysterectomy or ligation fallopian tube) or menopause for less than a year must have a negative urine test and be ready to use effective contraception (intrauterine device, hormonal contraceptive, condom, vaginal diaphragm with spermicide) through visit Day 22

Exclusion Criteria:

* Currently (within 2 weeks from the time of selection) with severe acute illness with or without fever.
* Participation in another therapy-related clinical trial within the past 3 months or plan to participate in a similar clinical trial at the same time it is.

Use any other vaccine for 4 weeks prior to joining or refusing to delay vaccination of such vaccines until after the visit on Day 22 (for groups ≥ 9 years) or day 49 (with groups <9 years old).

* Having been vaccinated against influenza in the past 11 months (only children 6 months to 8 years old who have been previously vaccinated with influenza vaccine (from birth) are also exclusion criteria).
* Use immunoglobulins or other hematological products within 3 months prior to study enrollment or plan to use these products prior to day 22 visit (for groups ≥ 9 years) or day 49 (with groups <9 years old).
* Suspected or certain acquired immunodeficiency.
* Long-term use (described as 14 consecutive days or more) immunosuppressants or other immunomodulatory therapies within 6 months prior to joining (for corticosteroids such as prednisone or substances similar to dose ≤ 0.5 mg / kg / day; topical steroids are allowed).
* Through historical exploitation or physical examination, there is an unstable disease, but according to the researcher's assessment, this may affect the implementation or the results of the study or increase the risk for the participants. researcher.
* Have experienced a previous hypersensitivity reaction after using any vaccine.
* Certain or suspected hypersensitivity reaction to any ingredient of the studied vaccine, including chicken protein or chicken eggs and rubber (from the rubber cap of the vaccine vial).
* Bleeding disorders or anticoagulant use within 3 weeks prior to selection. Have active TB or have symptoms of active tuberculosis, whatever the cause (self-reported).
* Are currently addicted to alcohol or using drugs that, according to researchers' assessment, could affect their ability to comply with research protocols.
* History of Guillain-Barré syndrome.
* Cancer or any malignant blood disease.
* Children under 1 year old but at birth with gestational age ≤ 36 and ≥ 43 weeks at birth and birthweight ≤ 2500g
* Children <60 months old with severe malnutrition aged II and above

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Experiencing Solicited Local and Systemic Adverse Events (AE) | Within 30 minutes of vaccination
  Solicited local and systemic AEs were assessed by study staff 30 minutes after vaccination.
Number of Subjects Experiencing Solicited Local and Systemic Adverse Events (AE) | within 7 days (day 1 to 7) of each vaccination
  Solicited local AEs were assessed by study staff 30 minutes after vaccination then daily for 7 days
Number of Subjects Experiencing Unsolicited Adverse Events (AE) | within 21 days (age group 9-17 and older than 60 years) or 49 days (group 6 months to 8 years) after each vaccination
  Unsolicited AEs were observed by study staff while the subject is at a clinic for a study visit or reported by the subject at any time. Any sign or symptom that would normally be considered a "solicited AE" (for example, fever, nausea, injection site pain) starting after 7 days post-vaccination was to be recorded as an unsolicited AE
Number of Subjects Experiencing Unsolicited Serious Adverse Events (SAE) | Day 1 to Day 91
  A serious adverse event (SAE) is defined as an AE that meets one of the following conditions:
  * Deadly.
  * Life-threatening.
  * Requires inpatient hospital admission or extended stay in hospital.
  * Causes birth defects.
  * Causes permanent or permanent injury or disability.
  * Critical medical events that may not be fatal, not life-threatening, or require inpatient treatment will be considered a SAE if it is judged by professional judgment that the incident would be potentially dangerous. subject's health and the need for medical or surgical intervention to prevent one of the aforementioned consequences
Number of Subjects With Seroconversion of Hemagglutination Inhibition (HAI) Antibodies for Vaccine Antigens, Overall and by Age Group | Day 22 (+7) for groups 9 years and above or 49 (+7) for groups of 6 months to under 9 years
  Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine

SECONDARY OUTCOMES:
Number of Subjects With Hemagglutination Inhibition (HAI) Antibody tiers ≥ 1:40 for each antigenic component of the vaccine | Day 22 or 49 after vaccination ( depending on age group)
  Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine
Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) Antibodies for Vaccine Antigens at Baseline and Day 22 or 49 after vaccination (depending on age group) for each antigenic component of the vaccine | Day 0, Day 22 and Day 49
  Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine
Geometric Mean Fold Change in HAI Antibody Titer, by Strain, Age Group, and Baseline Titer | Day 0, Day 22 and Day 49
  Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Pham N Hung, Prof., Principal Investigator — Vietnam Military Medical University
Locations (2):
- Vietnam (2):
  - CDC Ha Nam, Phủ Lý, Ha Nam
  - CDC Thai Binh, Thái Bình

IPD SHARING:
Plan to Share IPD: No